CLINICAL TRIAL: NCT05823571
Title: Phase 1a/1b Study of Itacitinib (INCB039110) for Cytokine Release Syndrome Prevention and Minimization of Immunosuppression Following Nonmyeloablative Related Partially HLA-mismatched Peripheral Blood Stem Cell Transplant (PBSCT) With High-dose Posttransplantation Cyclophosphamide in Older Patients (Age 60 Years)
Brief Title: Itacitinib With High-dose Posttransplantation Cyclophosphamide in Older Patients
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J2283; IRB00298829 (Other: JHMIRB)
Record Dates: First submitted 2023-04-10; First posted 2023-04-21 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Leukemia, Acute; Myelodysplastic Syndromes; Myelomonocytic Leukemia, Chronic; T-cell Prolymphocytic Leukemia; CML; Myeloproliferative Disorders; Multiple Myeloma; Plasma Cell Leukemia
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Leukemia, Prolymphocytic, T-Cell; Myeloproliferative Disorders; Multiple Myeloma; Leukemia, Plasma Cell | interventions — itacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Itacitinib (Experimental): Itacitinib will be given at 200 mg orally daily from day -3 to day 90. Itacitinib will be given in conjunction with one of four different regimens for immunosuppression. These 4 regimens are listed in Table 2, Section 5.2 of the protocol. Itacitinib may continue beyond day +90 if there is GVHD. NOTE: If patient develops GVHD requiring treatment after all immune suppression, including itacitinib, is stopped on day +90, the itacitinib will not be restarted and the patient will be treated per standard of care.
  Interventions: Drug: Itacitinib

INTERVENTIONS:
Drug: Itacitinib — A standard 3+3 design will be used to evaluate the safety of itacitinib plus different immunosuppression regimens. This study has four predefined Regimens that will be explored in the optimal Regimen-finding phase and are listed in Table 2 of the protocol. Itacitinib will be given in conjunction with each of four different regimens for immunosuppression. Regimen 1 is the current standard for our BMT patients, with a duration of MMF from day 5-35. Regimen 2 will decrease the duration of MMF from 35 to day 25. Regimen 3 will decrease the duration of MMF from 35 to day 15. Regimen 4 will eliminate MMF altogether. We will start with Regimen 1, which combines itacitinib with the current standard of immunosuppression. Progression through cohorts (Regimens) will be based on a standard 3+3 design to find the optimal regimen.

SUMMARY:
This research is being done to learn whether drug called itacitinib, which is a novel inflammation- and immune-lowering drug (immunosuppressant), can be given before and after non-myeloablative peripheral blood stem cell transplantation (PBSCT; also known as a 'mini' transplant) to help prevent certain complications such as cytokine release syndrome (CRS) for patients with blood cancers, using peripheral blood from a relative. The investigators will also examine if by using itacitinib the investigators can reduce the duration of MMF (other immune suppressive drug administration posttransplant).

DETAILED DESCRIPTION:
The NMA PBSC haplo transplant is associated with a higher risk of morbidity and mortality from the cytokine (IL-6 and others)-driven CRS and perhaps higher incidence of acute and chronic GVHD compared to bone marrow (BM) haplo allografting with post-transplant cyclophosphamide (PTCy). Notably, severe CRS (grade 3 and higher) appears to be more common in older patients (≥ 60 years) and is associated with significantly higher non-relapse mortality (NRM) in this patient group. Itacitinib has demonstrated safety, tolerability, ability to inhibit cytokines, including IL-6. Data also suggest that itacitinib can be administered safely in peri- and post-transplant period in the setting of Posttransplant CY immune prophylaxis and haploPBSCT with no evidence of delayed engraftment or delayed count recovery, with significant reduction in CRS compared to historical control, and a low rate of aGVHD, cGVHD, and NRM, and with no increase in relapse risk. Thus, the investigators propose a clinical study in which itacitinib will be used prophylactically in recipients age 60 years and older to prevent development of severe CRS, reduce severe CRS-associated NRM, and the incidence of severe GVHD, thus allowing further reduction in posttransplant immunosuppression therapy after PTCy-based NMA related partially-mismatched PB allografting.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a suitable related, HLA-haploidentical (partially mismatched) stem cell donor.
* Eligible diagnoses:

  1. Acute leukemias in complete remission with minimal residual disease
  2. Myelodysplastic syndrome (MDS) with at least one poor-risk feature
  3. Chronic myelomonocytic leukemia with at least one poor-risk feature
  4. T-cell PLL in PR or better prior to transplantation.
  5. Tyrosine kinase-refractory CML in first chronic phase, TKI-intolerant CML in first chronic phase, or CML in second or subsequent chronic phase.
  6. Philadelphia chromosome negative myeloproliferative disease (including myelofibrosis)
  7. Multiple myeloma or plasma cell leukemia with a PR or better to the last treatment regimen
* Age ≥ 60 years.
* Adequate end-organ function as measured by:

  1. Left ventricular ejection fraction ≥ 35% or shortening fraction > 25%
  2. Bilirubin ≤ 3.0 mg/dL (unless due to Gilbert's syndrome or hemolysis), and ALT and AST ≤ 5 x ULN
  3. FEV1 and FVC ≥ 40% of predicted
* ECOG performance status ≤ 2 or Karnofsky score ≥ 60

Exclusion Criteria:

* No active extramedullary leukemia or known active CNS involvement by malignancy.
* Any previous autologous HSCT must have occurred at least 3 months prior to start of conditioning.
* No previous allogeneic HSCT.
* Not pregnant or breast-feeding
* No uncontrolled infection.
* No known HIV infection.
* No active replicating HBV or HCV infection detected by PCR that requires treatment or at risk for HBV reactivation (positive HBsAg)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Number of participant deaths | 14 days
  Number of participant deaths will be used to assess the efficacy of itacitinib in preventing the occurrence of death.
Number of participants with grade 3 or higher CRS | 14 days
  Number of participants with grade 3 or higher CRS will be used to assess the efficacy of itacitinib in preventing the development of severe (grade 3 or higher) cytokine release syndrome (CRS).
Number of participants with grade 1-2 CRS that requires additional CRS-directed treatment | 14 days
  Number of participants with grade 1-2 CRS that requires additional CRS-directed treatment will be used to assess the efficacy of itacitinib in preventing the development of grade 1-2 CRS that requires additional CRS-directed treatment.
Number of participants with treatment limiting toxicities by Day 60 | 60 days
  Number of participants with treatment limiting toxicities by Day 60 will be used to identify the safe PTCy-based immunosuppressive regimen that incorporates itacitinib with tacrolimus and a reduced duration of immunosuppression with mycophenolate (MMF).

CONTACTS AND LOCATIONS:
Overall Officials: Ivana Gojo, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States